CLINICAL TRIAL: NCT00686231
Title: The Effect of Topical Administration of Nitroglycerin and Lidocaine Versus Lidocaine Alone of the Radial Artery Diameter
Brief Title: Radial Artery Dilation Study: The Effect of Topical Administration of Nitroglycerin and Lidocaine Versus Lidocaine Alone of the Radial Artery Diameter
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 56438-31921
Record Dates: First submitted 2008-05-19; First posted 2008-05-29 (Estimated); Results first posted 2010-07-22 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Healthy
Keywords: To determine if topical nitroglycerin acts to vasodilate the radial artery by a direct local action, or by systemic vasodilation; To determine if topical nitroglycerin dilates the radial artery in the presence of local anesthetic agents used in cardiac catheterization
MeSH Terms: interventions — Nitroglycerin; Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose Test 15mg NTG (Experimental): Nitroglycerin 15mg (NTG) applied topically to one wrist and placebo to the other wrist at Visit 1
  Interventions: Drug: Nitroglycerin 15mg; Drug: Placebo
- Dose Test 30mg NTG (Experimental): Nitroglycerin 30mg applied topically to one wrist and placebo to the other wrist at Visit 1
  Interventions: Drug: Nitroglycerin 30mg; Drug: Placebo
- Combination Test 20mg Lidocaine (Experimental): Lidocaine 20mg + Nitroglycerin 30mg applied topically to one wrist, Lidocaine 20mg + placebo applied to the other wrist, at Visit 2
  Interventions: Drug: Nitroglycerin 30mg; Drug: Lidocaine 20mg; Drug: Placebo
- Combination Test 40mg Lidocaine (Experimental): Lidocaine 40mg + Nitroglycerin 30mg applied topically to one wrist, Lidocaine 40mg + placebo applied to the other wrist, at Visit 2
  Interventions: Drug: Nitroglycerin 30mg; Drug: Lidocaine 40mg; Drug: Placebo

INTERVENTIONS:
Drug: Nitroglycerin 15mg — 15mg Nitroglycerin applied topically to one wrist
  Arms: Dose Test 15mg NTG
Drug: Nitroglycerin 30mg — 30mg Nitroglycerin applied topically to one wrist
  Arms: Combination Test 20mg Lidocaine; Combination Test 40mg Lidocaine; Dose Test 30mg NTG
Drug: Lidocaine 20mg — 20mg Lidocaine applied topically to one wrist in combination with nitroglycerin or placebo
  Arms: Combination Test 20mg Lidocaine
Drug: Lidocaine 40mg — 40mg Lidocaine applied topically to one wrist in combination with nitroglycerin or placebo
  Arms: Combination Test 40mg Lidocaine
Drug: Placebo — Topical skin moisturizing cream with same appearance as active agent
  Other Names: skin moisturizing cream

SUMMARY:
The radial artery, which is located on the outer side of the forearm, can be used in interventional procedures, such as cardiac catheterization, to provide access to the arterial blood supply. In order to facilitate successful catheterization of the artery, a dilated artery and one free of arterial spasm is desirable. The proposed study will randomize twenty three healthy subjects in 2 visits to determine the effect of topical nitroglycerin on radial artery vasodilation. Radial artery diameter will be measured with ultrasound at regular intervals up to two hours.

DETAILED DESCRIPTION:
During the first study visit, as a dose-optimizing study, each subject will be randomly assigned to one of two Dose-Test arms to receive either 15mg or 30mg of nitroglycerin on one wrist and placebo on the other. Radial artery diameter will be measured with ultrasound at regular intervals up to two hours. On the second study visit, the same participants will be randomly assigned to one of two Combination-Test arms to receive bilateral topical application of either 20mg or 40mg of lidocaine; the lidocaine will be applied in combination with 30mg of nitroglycerin on one wrist and in combination with placebo on the other wrist. Measurements of radial artery diameter will be performed as in the first visit.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent and comply with study requirements
* Patient who speak English

Exclusion Criteria:

* Presence or history of liver, cardiovascular, rheumatologic, cancer or renal disease.
* Current treatment with any vasodilator therapy
* Systolic blood pressure of less than 90 mmHg
* History of radial artery catheterization within the previous year
* Absence of radial artery blood flow in one or both arms
* Pregnancy.
* Active infection
* Staff members of the Cardiac Catheterization Laboratory.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2008-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF Medical Center, San Francisco, California, United States

REFERENCES:
- [Derived] Majure DT, Hallaux M, Yeghiazarians Y, Boyle AJ. Topical nitroglycerin and lidocaine locally vasodilate the radial artery without affecting systemic blood pressure: a dose-finding phase I study. J Crit Care. 2012 Oct;27(5):532.e9-13. doi: 10.1016/j.jcrc.2012.04.019. Epub 2012 Jun 12. PMID 22699036

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose-test 15mg: 15mg Nitroglycerin on one wrist and Placebo on the other
- Dose-test 30mg: 30mg Nitroglycerin on one wrist and Placebo on the other
- Combination Test 20mg: 30mg Nitroglycerin + 20mg Lidocaine on one wrist, and Placebo + 20mg Lidocaine on the other wrist
- Combination Test 40mg: 30mg Nitroglycerin + 40mg Lidocaine on one wrist, and Placebo + 40mg Lidocaine on the other
Period: Dose Test - Visit 1
Arm/Group | Dose-test 15mg | Dose-test 30mg | Combination Test 20mg | Combination Test 40mg
Started | 12 | 7 | 0 | 0
Completed | 12 | 7 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Combination Test - Visit 2
Arm/Group | Dose-test 15mg | Dose-test 30mg | Combination Test 20mg | Combination Test 40mg
Started | 0 | 0 | 10 | 9
Completed | 0 | 0 | 10 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The PI has left the institution and all efforts to locate per arm data for this module have been exhausted and therefore cannot be reported.
Groups:
- Overall Study: Healthy subjects older than 18 years were recruited and randomly assigned to one of two study arms on each of two separate study visits. Visit 1: 15mg Nitroglycerin vs. 30 mg Nitroglycerin on one wrist and placebo on the other wrist. Visit 2: 20mg Lidocaine vs. 40mg Lidocaine in combination with Nitroglycerin on one wrist and with placebo on the other wrist.
Arm/Group | Overall Study
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Diameter of Radial Artery as a Dose Test for Nitroglycerin
Description: Radial artery diameter was measured with ultrasonography using a high-frequency (13 MHz) linear array transducer 2 cm proximal to the radial styloid process.
Time Frame: Baseline, 10 minutes, 30 minutes, 60 minutes, and 120 minutes after topical application at Visit 1
Population: 19 participants were randomized to receive 15mg (n=12) or 30mg (n=7) nitroglycerin on one wrist, and placebo on the other
Measure: Mean (Standard Deviation); unit: percent diameter change
Units Other Than Participants: radial artery (wrist)
Groups:
- Placebo: Moisturizing skin cream as a matching placebo was topically applied to one wrist, where 15mg or 30mg (by random assignment) Nitroglycerin was applied to the other wrist
- 15mg Nitroglycerin: 15mg of nitroglycerin was administered topically on one wrist (where matching placebo was applied to the other wrist)
- 30mg Nitroglycerin: 30mg of nitroglycerin was administered topically on one wrist (where matching placebo was applied to the other wrist)
Arm/Group | Placebo | 15mg Nitroglycerin | 30mg Nitroglycerin
Number analyzed (Participants) | 19 | 12 | 7
Number analyzed (radial artery (wrist)) | 19 | 12 | 7
percent diameter change
  10 minutes | -0.8 (0.5) | -0.2 (2.8) | 6.4 (4.5)
  30 minutes | 2.5 (12.5) | 0.8 (3.5) | 14.9 (18.1)
  60 minutes | 3.3 (6.5) | 10.2 (5.4) | 21.5 (6.6)
  120 minutes | 5.9 (6.5) | 8.8 (10.1) | 28.5 (12.1)

2. Primary Outcome: Percent Change From Baseline in Radial Artery Diameter to Compare Combination of Nitroglycerin or Placebo and Lidocaine (20mg or 40mg)
Description: Radial artery diameter was measured with ultrasonography using a high-frequency (13 MHz) linear array transducer 2 cm proximal to the radial styloid process. To compare combination of (Lidocaine + Nitroglycerin) or (Lidocaine + placebo), at visit 2, participants randomized to Comparison A received 30mg NTG + 20mg Lidocaine on one wrist, and placebo + 20mg Lidocaine on the other wrist; participants randomized to Comparison B received 30mg Nitroglycerin + 40mg Lidocaine on one wrist, and placebo + 40mg Lidocaine on the other wrist.
Time Frame: Baseline, 10 minutes, 30 minutes, 60 minutes, and 120 minutes after topical application at Visit 2
Population: 10 participants (20 wrists) received 30mg NTG + 20mg Lidocaine on one wrist, and placebo + 20mg Lidocaine on the other wrist; 9 participants (18 wrists) received 30mg NTG + 40mg Lidocaine on one wrist, and placebo + 40mg Lidocaine on the other wrist.
Measure: Mean (Standard Deviation); unit: percent diameter change
Units Other Than Participants: Radial Artery
Groups:
- Lidocaine 20mg + Placebo: 20mg combination test: lidocaine + placebo
- Lidocaine 20mg + Nitroglycerin 30mg: 20mg combination test: lidocaine + nitroglycerin
- Lidocaine 40mg + Placebo: 40mg combination test: lidocaine + placebo
- Lidocaine 40mg + Nitroglycerin 30mg: 40mg combination test: lidocaine + nitroglycerin
Arm/Group | Lidocaine 20mg + Placebo | Lidocaine 20mg + Nitroglycerin 30mg | Lidocaine 40mg + Placebo | Lidocaine 40mg + Nitroglycerin 30mg
Number analyzed (Participants) | 10 | 10 | 9 | 9
Number analyzed (Radial Artery) | 10 | 10 | 9 | 9
percent diameter change
  10 minutes | 4 (3.6) | 4.9 (7.2) | 1.6 (3.0) | 3.4 (3.0)
  30 minutes | 5.3 (5.8) | 11.0 (10.6) | 2.9 (1.8) | 10.6 (6.5)
  60 minutes | 8.4 (7.4) | 18.2 (9.4) | 2.5 (3.2) | 17.2 (9.2)
  120 minutes | 5.7 (6.8) | 18.5 (8.7) | 4.1 (3.9) | 22.1 (12.0)

ADVERSE EVENTS:
Groups:
- Study: Healthy subjects older than 18 years were recruited and randomly assigned to one of two study arms on each of two separate study visits. Visit 1: 15mg Nitroglycerin vs. 30 mg Nitroglycerin on one wrist and placebo on the other wrist. Visit 2: 20mg Lidocaine vs. 40mg Lidocaine in combination with Nitroglycerin on one wrist and with placebo on the other wrist.
Arm/Group | Study
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes